CLINICAL TRIAL: NCT00575718
Title: Presurgical Smoking Cessation Intervention for Cancer Patients: The Resolve Study
Brief Title: Smoking Cessation Intervention for Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02-094
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Newly Diagnosed Cancer Patients
Keywords: Quitting tobacco; tobacco use
MeSH Terms: conditions — Tobacco Use | interventions — Nicotine Replacement Therapy

ARMS (2):
- 1 (Active Comparator): Hospital Counseling + Nicotine Replacement Therapy (HC+NRT)
  Interventions: Behavioral: Hospital Counseling + Nicotine Replacement Therapy. questionaires
- 2 (Experimental): Hospital Counseling + Nicotine Replacement Therapy + Pre-surgical Schedule Reduced Smoking (HC+NRT+PS/SRS)
  Interventions: Behavioral: Hospital Counseling + Nicotine Replacement + Presurgical Scheduled Reduced Smoking, questionaires

INTERVENTIONS:
Behavioral: Hospital Counseling + Nicotine Replacement Therapy. questionaires — brief face-to-face or telephone tobacco cessation counseling provided by a tobacco cessation specialist prior to admission and during hospitalization (15-20 minutes per encounter)provision of multi-media self-help materials (e.g., "Smoking Cessation Guide for Cancer Patients and Their Families") tailored to address cancer-specific issues such as the benefits and barriers of quitting for cancer patients; 3) tobacco cessation pharmacotherapy, unless medically contraindicated (for this study we will standardize the pharmacotherapy as transdermal nicotine patch), and; 4) two brief telephone counseling (15 minutes) sessions completed as seen clinically appropriate by the tobacco cessation specialists. The content of these counseling sessions is based on the patient's smoking status.
  Arms: 1
Behavioral: Hospital Counseling + Nicotine Replacement + Presurgical Scheduled Reduced Smoking, questionaires — Same components of HC+NRT as well as the PS/SRS enhancement.The research team will provide education about scheduled reduced smoking either in person or over the phone. Purpose of the training session, will be audio taped, to prepare participants for daily PDA use over the dur of the scheduled-reduced smoking intervention. Training will demonstrate use of PDA and simulate common technical and procedural issues that might arise during the intervention (e.g., forgetting to record a cigarette or wake time; repeating a day's schedule if needed, prior to the quit date). The simulation will reflect anticipated problems and those identified by users of the PDA. A study helpline number and instructional manual will be provided. A member of the research staff will contact the study participants, once the reduced smoking schedule has begun, to check that the patient understands the schedule and that the PDA is working properly. Estimate patient training with the PDA will require 30 minutes.
  Arms: 2

SUMMARY:
The purpose of this study is to see if we can find ways to improve the treatment of tobacco dependence in patients who have cancer or may have cancer. We will compare two ways to help people quit tobacco use before surgery and to stay quit after surgery. One way is a scheduled reduced smoking program followed by use of the nicotine patch. In this program, the tobacco user will gradually cut down on their tobacco use until they quit. Once they quit, they will be offered the nicotine patch. We will compare this approach to our current program of counseling and use of nicotine patch. What we learn from this study may help us to develop new ways to help tobacco users and improve our current smoking cessation program.

DETAILED DESCRIPTION:
Smoking cessation offers an important way for newly diagnosed cancer patients to take an active role in their treatment and recovery. Quitting tobacco use decreases cancer patients' risk of disease recurrence and development of second primary cancers. In addition, preoperative tobacco cessation may reduce the likelihood of perioperative pulmonary, cardiovascular, and wound healing complications. Due to increased awareness of the health hazards of tobacco use, rates of cessation after cancer diagnosis are high. However, 35% to 69% of patients continue to use tobacco and this is largely due to strong barriers to quitting (low-self efficacy, psychological distress) rather than lack of positive intentions to quit. Previous attempts to increase smoking cessation among the medically ill have provided intervention either during or after hospitalization.

We propose that the period immediately prior to hospitalization and surgery represents a unique window of opportunity, or "teachable moment," for smoking cessation that could take full advantage of patients' enhanced health awareness and quitting motivation, strong physician quitting advice, and patients' heightened desire to take an active role in their care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Smokers who typically smoke > 8 cigarettes per day who have smoked within the last 7 days or other tobacco users with high frequency of use (> 8 per day) within the last 7 days;
* Diagnosed with cancer or have a mass suspicious of cancer that is NOT distant metastatic cancer at the time of enrollment;
* Likely candidate for surgical treatment no sooner than 7 days from study entry;
* Absence of gross psychopathology or cognitive impairment;
* Can be reached by telephone;
* Have manual dexterity and sensory (i.e., visual and auditory) acuity sufficient to use a Personal Digital Assistant (PDA);
* Provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2002-10-22 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
efficacy of a presurgical smoking cessation intervention that adds scheduled reduced smoking, a highly effective behavioral treatment in non-medically ill tobacco users, to enhanced usual care, i.e., hospital counseling and nicotine replacement therapy. | will be measured at hospital admission, and 3 and 6 months post-hospital admission.

SECONDARY OUTCOMES:
whether addition of a presurgical scheduled reduced smoking intervention improves smoking cessation and long-term abstinence rates c/w hospital counseling and nicotine transdermal patch (enhanced usual care) for recently diagnosed cancer patients. | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org